CLINICAL TRIAL: NCT00353041
Title: A Study of the Effect of Time on Topical Anesthetic Efficacy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: UToronto
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2006-07-17 (Estimated); Status verified 2006-07

CONDITIONS: Pain
Keywords: topical; anesthetic; pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

INTERVENTIONS:
Drug: lidocaine topical

SUMMARY:
This is a study of the effect of time on the effectiveness of topical anesthetics in the mouth. The Null Hypothesis is: Regardless of the time of application over a 10-minute period, there is no difference in the clinical effectiveness of the topical anesthetic 5% lidocaine on (a) the pain of needle stick insertion and (b) the pain of local anaesthetic administration.

DETAILED DESCRIPTION:
The study design will be a double blind randomized controlled split-mouth clinical trial. It is proposed to compare the effectiveness of the standard topical anesthetic 5% lidocaine with a placebo over the time period of 2, 5 and 10 minutes after application. The topical will be placed on the palatal soft tissue where the perception of pain is the highest in the oral cavity. Both the pain of needle insertion and the pain of local anesthetic injection will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. In good health (ASA 1 or ASA 2)
2. Weight between 40-100kg, inclusive.
3. Between ages 18-70, inclusive.
4. Informed consent

Exclusion Criteria:

1. ASA 3 or higher.
2. History of allergy to sulfites, lidocaine or mepivacaine.
3. Taking any analgesic 48hrs before testing, such as an NSAID, opioid, or acetaminophen.
4. Pregnancy.
5. Recent oral trauma.
6. Lack of informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2006-07; Study Completion 2006-12

PRIMARY OUTCOMES:
pain

SECONDARY OUTCOMES:
Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Haas, DDS, PhD, Principal Investigator — University of Toronto
Locations (1):
- Faculty of Dentistry, Toronto, Ontario, Canada